Consent to participate in non-biomedical research: Babies' Expectations about Racial Interactions

Study researchers led by Professor Amanda Woodward at University of Chicago are running this study, "Babies' Expectations about Racial Interactions," on Lookit.

## Purpose

At the Infant Learning and Development Laboratory at the University of Chicago, we are interested in how infants and young children reason about the world and how they learn from their interactions with other people. Through our research, we hope to better understand children's early reasoning, and how that thinking changes as they grow older, in order to paint a clearer picture of development for scientists, parents and educators. In today's study, we are investigating how social categories (such as race and language groups) and social experiences affect children's learning. Our goal in these studies is to see what children naturally do in response to seeing people interact and whether they pay attention to the person's race when processing these interactions. Please understand that there are no right or wrong answers. Our findings do not allow us to draw meaningful conclusions about an individual child's abilities, although they can provide information about general patterns in infant development.

#### **Procedures**

This study takes about 15 minutes to complete. Your child will be shown videos of two people. There will be three types of videos: (1) two people talking; (2) two people saying hi; and (3) two people turning their backs to each other. We are interested in what babies think about people and their interactions according to the race of the people they saw. We will ask you (the parent) to turn around, close your eyes, or look down to avoid influencing your child's responses. There are no anticipated risks associated with participating. To better understand your child's social environment, we will also ask you to fill out a questionnaire after the experiment and an additional survey about the people your child interacts with regularly.

#### Participation

You and your child are free to choose whether to be in this study. If you and your child choose to participate, it's okay to stop at any point during the session. Please do pause or stop the session if your child becomes very fussy or does not want to participate! If this is a study with multiple sessions, it's okay not to complete all the sessions.

### Payment

After you finish the study, we will email you a \$5 gift card within the next week. In addition, you can earn an additional \$5 gift card if you fill out another external survey linked at the end of the study. To be eligible for the gift card your child must be in the age range for this study, you need to submit a valid consent statement, and we need to see that there is a child with you. But we will send a gift card even if you do not finish the whole study or we are not able to use your child's data! There are no other direct benefits to you or your child from participating, but we hope you will enjoy the experience.

#### Data collection and webcam recording

During the session, you and your child will be recorded via your computer's webcam and microphone. Video recordings and other data you enter are sent securely to our lab. At the end of the session, you will be prompted to choose a privacy level for your webcam recordings. You will have the option to withdraw your video data at this point.

Data is stored securely on Lookit servers and by researchers. However, there is always a small risk that data transmitted over the internet may be intercepted or that the security of stored data may be compromised.

No video clips will be published or shared unless you allow this when selecting a privacy level. If we do not receive a consent recording (the video you'll make to the right) for this session and cannot verify that you agreed to participate, no other video from your session will be viewed.

# Use of data by study researchers

The research group led by Professor Amanda Woodward at University of Chicago will have access to video and other data collected during this session. We will also have access to your account profile, demographic survey, and the child profile for the child who is participating, including changes you make in the future to any of this information. We may study your child's responses in connection with his or her previous responses to this or other studies run by our group, or demographic survey responses.

Trained research assistants will view these videos to measure how long infants looked. These research assistants will not have access to identifying information, including name and birthdate, when they are coding these videos. We will not report any identifying information in order to maintain confidentiality. This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents or data that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding. The Certificate of Confidentiality will not be used to prevent disclosures for any purpose you have consented to in this informed consent document, such as the sharing of videos or pictures of your child. The Certificate of Confidentiality will also not be used to prevent disclosure of child abuse or neglect as required by federal, state, or local law.

## Use of data by Lookit

Because this study is being run on the Lookit platform, researchers working on the Lookit project at MIT will also have access to the data collected during this session, in addition to your account data, child profiles, and demographic survey responses. This data may be used by Lookit to detect and fix technical problems or identify new features that would be helpful; provide support to study researchers; assess data quality (for instance, how well an observer can tell which direction children are looking); evaluate the site's success in reaching a diverse population; and characterize family engagement (for instance, looking at what aspects of a study make parents more interested in coming back later).

### Publication of results

The results of the research may be presented at scientific meetings or published in scientific journals. Raw data (for instance, looking times to the left and right of the screen) may be published when it cannot identify children. We never publish children's

birthdates or names, and we never publish your demographic data in conjunction with your child's video.

# Researcher contact information

This study is run by Professor Amanda Woodward at University of Chicago. If you or your child have any questions or concerns about this study, or in the very unlikely event of a research-related injury, please contact woodward@uchicago.edu.

If you or your child have any questions or concerns about the Lookit platform, please contact Kim Scott at kimscott@mit.edu or 617 324 4859.